CLINICAL TRIAL: NCT00028782
Title: The Detection of Tumor Hypoxia and Vascularity in Patients Undergoing Intraperitoneal Photodynamic Therapy
Brief Title: EF5 in Detecting Oxygen Level and Blood Vessels in Tumor Cells of Patients Undergoing Photodynamic Therapy for Intraperitoneal or Pleural Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2012-02438; UPCC# 05901; P01CA087971 (NIH); CDR0000069134 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Malignant Mesothelioma; Localized Malignant Mesothelioma; Malignant Ascites; Primary Peritoneal Cavity Cancer; Recurrent Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Etanidazole

ARMS (1):
- Diagnostic (etanidazole) (Experimental): Patients receive etanidazole derivative EF5 IV over 1-2 hours. Approximately 48 hours after EF5 administration, patients with intraperitoneal tumors undergo surgical resection. Patients with pleural tumors undergo surgical resection approximately 24 hours after EF5 administration. Tumors are then analyzed for EF5 binding and microvascular density by immunohistochemistry and fluorescent antibody techniques.
  Interventions: Drug: etanidazole; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: etanidazole — Given IV
  Other Names: 2-nitro-imidazole derivative; SR-2508
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well EF5 works in detecting oxygen level and blood vessels in tumor cells of patients who are undergoing photodynamic therapy for intraperitoneal or pleural cancer. Diagnostic procedures using EF5 to detect oxygen level and blood vessels in tumor cells may help to improve the way photodynamic therapy is given

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the level of hypoxia through etanidazole derivative EF5 binding in patients with intraperitoneal or pleural malignancies treated with photodynamic therapy.

II. Determine the microvascular density in this patient population. III. Determine the relationships between levels of hypoxia, measures of microvascular density, and photosensitizer levels in this patient population.

IV. Correlate hypoxia and photosensitizer levels with clinical outcome in this patient population.

V. Determine the toxic effects of EF5 in this patient population.

OUTLINE: This is a multicenter study.

Patients receive etanidazole derivative EF5 IV over 1-2 hours. Approximately 48 hours after EF5 administration, patients with intraperitoneal tumors undergo surgical resection. Patients with pleural tumors undergo surgical resection approximately 24 hours after EF5 administration. Tumors are then analyzed for EF5 binding and microvascular density by immunohistochemistry and fluorescent antibody techniques.

Patients are followed at 2 weeks and at 30-45 days post EF5 infusion.

PROJECTED ACCRUAL: A total of 80 patients (50 with intraperitoneal malignancy and 30 with pleural malignancy) will be accrued for this study within 2.5 years. Patients are stratified by disease (intraperitoneal malignancy vs pleural malignancy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intraperitoneal or pleural malignancy
* Currently enrolled on 1 of 3 photodynamic therapy trials (UPCC-2997, UPCC-4997, or UPCC-05503)

  * Plan to undergo surgery for treatment on one of these protocols
* Patients with suspected recurrent disease undergoing surgery for diagnosis and debulking allowed if frozen section shows malignant disease
* No active extra-abdominal metastatic disease and/or intrahepatic involvement secondary to metastatic carcinoma
* No borderline tumors of low malignant potential
* No abdominal disease that cannot be debulked to less than 5 mm residual disease in maximal dimension
* Performance status - ECOG 0-2
* WBC at least 2,000/mm^3
* Platelet count greater than 100,000/mm^3
* Bilirubin less than 1.5 mg/dL
* No severe liver disease
* No cirrhosis
* No grade III or IV elevations in liver function studies
* Creatinine no greater than upper limit of normal
* Creatinine clearance at least 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study treatment
* Weight no more than 130 kg
* HIV negative
* Able to tolerate anesthesia or major surgery
* No grade III or IV peripheral neuropathy
* No regional enteritis or ulcerative colitis
* No contraindication for anesthesia or major surgery
* Prior combination chemotherapy for malignancy allowed
* No concurrent chemotherapy except for recurrent or persistent disease
* No concurrent radiotherapy except for recurrent or persistent disease
* Prior surgery for malignancy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-10; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Level of hypoxia in tumor nodules | At the completion of surgery
  Exploratory techniques will be used to describe patterns of EF5 binding as well as MVD within and among patients.
Inter- and intra-patient variability of hypoxia by EF5 binding | At the completion of surgery
  Inter- and intra-subject variability can be estimated using summary statistics (standard deviations, or the range of data).
Levels of microvascular density by PECAM/CD31 staining | At the completion of surgery
  Distributions of the four EF5 binding variables and MVD will be examined graphically we anticipate that certain variables may have a Poisson distribution.
Relationships among levels of hypoxia, microvascular density, and photosensitizer levels | At the completion of surgery
Associations between hypoxia and photosensitizer levels in tumor nodules with clinical outcome periodically until disease recurrence | Not Provided

SECONDARY OUTCOMES:
Toxicity of EF5 administration | Up to 45 days after EF5 infusion
  All observed toxicities will be graded, tabled for each stratum (IP study) and for the entire study and summarized by frequencies and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States